CLINICAL TRIAL: NCT07250867
Title: Safety and Efficacy of Lidocaine Versus Ketamine Infusion or Both Together as a Treatment Modality in Patient With Resistant Orofacial Pain; Double Blinded Randomized Study.
Brief Title: Safety and Efficacy of Lidocaine Versus Ketamine Infusion for Resistant Orofacial Pain
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed mustafa ahmed, Resident in Anesthesia, Intensive Care, and Pain Management Department, Faculty of Medicine, Assiut University., Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Lidocaine versus Ketamine
Record Dates: First submitted 2025-11-19; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Orofacial Pain
Keywords: Orofacial Pain
MeSH Terms: conditions — Facial Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lidocaine Infusion Group (Experimental)
  Interventions: Drug: Lidocaine Intravenous Infusion
- Ketamine Infusion Group (Experimental)
  Interventions: Drug: Ketamine intravenous infusion
- Lidocaine-Ketamine Combination Group (Experimental)
  Interventions: Drug: Combined lidocaine and ketamine intravenous infusion

INTERVENTIONS:
Drug: Lidocaine Intravenous Infusion — Participants receive a slow intravenous infusion of lidocaine at a dose of 5 mg/kg (not exceeding 500 mg in total), diluted in 0.9% saline and administered over a 4-hour period, once weekly for three consecutive weeks. Continuous monitoring of cardiovascular and neurological status is provided during and after infusion to assess for efficacy and safety in cases of treatment-resistant orofacial pain.
  Arms: Lidocaine Infusion Group
Drug: Ketamine intravenous infusion — Participants receive a slow intravenous infusion of ketamine at a dose of 0.3 mg/kg, diluted in 0.9% saline and delivered over 4 hours, once weekly for three consecutive weeks. The procedure includes monitoring for cardiovascular and CNS adverse effects. This intervention aims to evaluate the analgesic and safety profile of ketamine in patients with persistent orofacial pain unresponsive to standard therapies.
  Arms: Ketamine Infusion Group
Drug: Combined lidocaine and ketamine intravenous infusion — Participants receive a single intravenous infusion containing both lidocaine (2.5 mg/kg) and ketamine (0.15 mg/kg) diluted in 0.9% saline, administered over 4 hours, once weekly for three consecutive weeks. This intervention is designed to determine whether the combination of lidocaine and ketamine provides synergistic analgesic effects and improved tolerability compared to either drug alone in treating resistant orofacial pain.
  Arms: Lidocaine-Ketamine Combination Group

SUMMARY:
A prospective, randomized, double-blind clinical trial comparing the safety and efficacy of intravenous lidocaine, ketamine, and their combination as treatment options for patients suffering from treatment-resistant orofacial pain. The study measures pain reduction primarily using the Visual Analog Scale and evaluates safety and tolerability over a follow-up period of 6 months.

DETAILED DESCRIPTION:
This study aims to assess and compare the analgesic efficacy and safety profiles of intravenous lidocaine, ketamine, and a combined infusion of both in adult patients with orofacial pain that is resistant to conventional medical or interventional therapies. Using a randomized, double-blind design, 105 patients will be allocated equally into three parallel groups receiving either lidocaine infusion (5 mg/kg over 4 hours), ketamine infusion (0.3 mg/kg over 4 hours), or a combination infusion of lidocaine (2.5 mg/kg) and ketamine (0.15 mg/kg) over 3 consecutive weeks. Primary efficacy will be assessed by changes in pain intensity measured by the Visual Analog Scale (VAS) from baseline through follow-up visits at the 2nd and 3rd infusions, and 1, 3, and 6 months post-treatment. Secondary outcomes include cortisol level changes, depression assessment via PLAT-Q, and adverse events monitored during and after infusions. Strict inclusion and exclusion criteria will ensure patient safety and reliability of results. Data will be analyzed using one-way ANOVA and repeated measures ANOVA for continuous variables with significance set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

- Adults aged > 18 years

Resistant orofacial pain patients with failed medical or interventional treatment

Diagnosed with one or more of the following:

Trigeminal neuralgia

Temporomandibular joint (TMJ) dysfunction

Malignant otitis externa

Migraine

Atypical facial pain

Exclusion Criteria:

- Debilitating cardiac disease

Uncontrolled hypertension

Known allergies to lidocaine or ketamine

Severe renal or hepatic impairment

Pregnancy or breastfeeding

History of substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Analog Scale (VAS) Pain Score | Baseline, prior to 2nd infusion, prior to 3rd infusion, 1 month, 3 months, and 6 months after intervention
  Reduction in pain intensity as measured using the Visual Analog Scale (VAS), a 0-10 scale where 0 represents no pain and 10 represents the worst pain imaginable. The VAS will be assessed at baseline (before the first infusion) and at each follow-up visit (prior to 2nd infusion, prior to 3rd infusion, 1 month, 3 months, and 6 months after the intervention) to determine the effect of each treatment on resistant orofacial pain.